CLINICAL TRIAL: NCT04013347
Title: Evaluation of Anatomopathological, Oncological and Surgical Outcomes in Relation to the Different Times Between the End of Neoadjuvant Treatment and Surgery
Brief Title: Outcomes of Resection at Different Times Between the End of Neoadjuvant Treatment and Surgery
Status: Completed | Type: Observational
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Vincenzo La Vaccara, Principal Investigator, Campus Bio-Medico University
Other Study IDs: 08/17 OSS ComEt CBM
Record Dates: First submitted 2019-06-28; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Neoadjuvant Chemoradiotherapy; Rectal Tumor; Surgery; Surgery--Complications
MeSH Terms: conditions — Rectal Neoplasms | interventions — Proctectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Early Surgery: Surgery after ≤ 42 days from the end of neoadjuvant radio-chemotherapy
  Interventions: Procedure: Rectal Resection
- Late Surgery: Surgery after 43-56 days from the end of neoadjuvant radio-chemotherapy
  Interventions: Procedure: Rectal Resection
- Very Late Surgery: Surgery after 57 or more days from the end of neoadjuvant radio-chemotherapy
  Interventions: Procedure: Rectal Resection

INTERVENTIONS:
Procedure: Rectal Resection — Low Anterior Resection and Abdominoperineal Resection

SUMMARY:
Neoadjuvant radio-chemotherapy (NRCT) represents a milestone in the treatment of selected rectal tumours. Ideal time interval between the end of NRCT and surgery is still debated; a 6-8 weeks time interval is considered optimal, but shorter or longer intervals have been associated with better oncological outcomes. Moreover, there is a lack of data about clinical postoperative outcomes and different time intervals after the end of NRCT. Here, effect that different time intervals have on postoperative complications with particular regard to the anastomotic dehiscence have been evaluated.

Methods One hundred-sixty-seven patients underwent surgery after long-course NRCT. Three different time intervals were considered: (0-42; 43-56; >57 days).

DETAILED DESCRIPTION:
Neoadjuvant radio-chemotherapy (NRCT) represents a milestone in the treatment of selected rectal adenocarcinoma. Even though a 6-8 weeks' time interval after the end of NRCT and surgery is considered ideal, the optimal time for surgery is still controversial.

ELIGIBILITY:
Inclusion Criteria:

- patients with rectal adenocarcinoma who underwent to resection after combined NRCT at University Campus Bio-Medico di Roma from January 2005 to March 2015.

To evaluate the anastomotic dehiscence were excluded patients undergone to Abdomino-perineal resection (APR) and 4 patients for whom data were not available.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One hundred and sixty-seven patients with rectal adenocarcinoma who underwent to resection after combined NRCT at University Campus Bio-Medico di Roma from January 2005 to March 2015 were retrospectively analysed.
Sampling Method: Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2017-03-21 (Actual)

PRIMARY OUTCOMES:
number of patient with low tumor regression grade | 1 week after surgery
  rate of low tumor regression grade (1-2)
number of patient with surgical complications | 1 month after surgery
  rate of surgical complications

SECONDARY OUTCOMES:
number of patient with anastomotic dehiscence | 1 month after surgery
  rate of anastomotic dehiscence

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caputo D, Angeletti S, Fiore M, Ciccozzi M, Coppola A, Cartillone M, La Vaccara V, Spagnolo G, Trodella L, Coppola R. Delayed surgery after radio-chemotherapy for rectal adenocarcinoma is protective for anastomotic dehiscence: a single-center observational retrospective cohort study. Updates Surg. 2020 Jun;72(2):469-475. doi: 10.1007/s13304-020-00770-1. Epub 2020 Apr 18. PMID 32306273